CLINICAL TRIAL: NCT02202265
Title: Effect of Polymorphisms in CD36 and STAT3 Genes on Different Dietary Interventions Among Patients With Coronary Artery Disease: a Randomized Clinical Trial With a Nutrigenetic Approach
Brief Title: Polymorphisms in CD36 and STAT3 Genes and Different Dietary Interventions Among Patients With Coronary Artery Disease
Acronym: GENUTRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 48612013
Record Dates: First submitted 2014-07-18; First posted 2014-07-28 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease
Keywords: Heart Diseases
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases | interventions — Olive Oil; Nuts

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control diet (standard dietary) (Active Comparator): Patients will receive a control diet based on standard dietary guidelines
  Interventions: Dietary Supplement: Control diet
- Olive oil (30ml a day) (Experimental): Patients will receive a control diet based on standard dietary guidelines + 30ml of olive oil a day
  Interventions: Dietary Supplement: Olive oil
- Nuts (30g a day) (Experimental): Patients will receive a control diet based on standard dietary guidelines plus 30g of nuts a day
  Interventions: Dietary Supplement: Nuts

INTERVENTIONS:
Dietary Supplement: Olive oil — 30ml a day of olive oil
  Arms: Olive oil (30ml a day)
Dietary Supplement: Nuts — 30g a day of nuts
  Arms: Nuts (30g a day)
Dietary Supplement: Control diet — Diet based on standard guidelines
  Arms: Control diet (standard dietary)

SUMMARY:
Background: Cardiovascular diseases are the major health problem worldwide and the understanding of genetic contributions on the development of cardiovascular diseases is increasing significantly. The CD36 is a protein associated with uptake of oxidized forms of LDL and the single nucleotide polymorphism (SNP) rs1761667 A/G in the CD36 gene is correlated with increased consumption of total fat. The transcription factor STAT3 is released during the inflammatory acute phase response and the SNP rs8069645 G/A in the STAT3 gene is associated with abdominal obesity and higher intake of saturated fat. Studies have been shown the benefits of the Mediterranean diet in secondary prevention of cardiovascular disease and these dietary patterns have been often studied with nutrigenetic approach; these studies, however, are often limited to European populations, making it difficult to generalize to different populations.

Hypothesis: Different dietary approaches may similarly influence in modifying metabolic, inflammatory and anthropometric profile, especially among patients with coronary arterial disease (CAD). The genetic interaction with environmental factors such as the nutrient intake, and the prescription of a different diet according to individual genotype, could influence the development and/or the treatment of cardiovascular diseases.

Objective: To evaluate the effect of three dietary approaches on metabolic, inflammatory and anthropometric profile in patients with CAD and possible interactions with polymorphisms in CD36 and STAT3 genes.

DETAILED DESCRIPTION:
A randomized clinical trial with a nutrigenetic approach among patients ≥ 40 years diagnosed with CAD. Randomization will be made in blocks from a list of random numbers generated by site www.randomization.org (sealed opaque envelopes). A questionnaire with demographic and clinical data will be applied; systolic and diastolic blood pressure, waist, hip and neck circumferences, height and weight will be assessed. Nutrients intake will be assessed through a food diary. Laboratory evaluation will consist of lipid profile (LDL-cholesterol, HDL-cholesterol and total cholesterol, serum triglycerides), glycemic profile (fasting plasma glucose, glycated hemoglobin) and inflammatory profile (high-sensitivity C-reactive protein, fibrinogen, TNF-alpha, interleukin-6 and interleukin-10). Genotyping will be made by TaqMan SNP Genotyping Assay®. Patients will be randomized in three groups: Group 1 Intervention [Supplementation with nuts (SN)]: standard dietary guidelines + 30g of nuts a day; Group 2 Intervention [Supplementation with olive oil (SAO)]: standard dietary guidelines + 30ml of olive oil a day; Group 3 [Control diet (CO)]: standard dietary guidelines. Patients will be followed for three months (12 weeks) and the primary endpoint will be the change in LDL-cholesterol. The follow-up visits will be made at 30 days, 60 days and 90 days (final visit).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with coronary arterial disease.

Exclusion Criteria:

* Psychiatric disease;
* Morbid obesity (BMI ≥ 40mg/m2);
* Expectancy of life less than 6 months;
* Pregnancy or lactation;
* Renal failure (in dialysis);
* Congestive heart failure;
* Prior organ transplantation;
* Patients in wheelchair;
* Use of vitamin/nutritional supplements;
* Chronic use of non steroidal anti-inflammatory drugs;
* Participation in another experimental study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-06-17 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
LDL | twelve weeks
  LDL-cholesterol, in mg/dL

SECONDARY OUTCOMES:
TC | twelve weeks
  total cholesterol (TC), in mg/dL)
NHDL | twelve weeks
  non-HDL-cholesterol, in mg/dL
HDL | twelve weeks
  HDL-cholesterol, in mg/dL
TG | twelve weeks
  serum triglyceride, in mg/dL
TyG index | twelve weeks
  Triglycerides/fasting glucose index, calculated according to (fasting triglycerides [mg/dL] x fasting glucose [mg/dL])/2
HbA1C | twelve weeks
  glycated hemoglobin (HbA1C), in %
FG | twelve weeks
  fasting glucose, in mg/dL
Insulin | twelve weeks
  serum insulin, in UI/mL
HOMA-IR | twelve weeks
  Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), calculated according to fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5
inflammatory profile | twelve weeks
  CRP-us, in mg/dL; IL-6, in mg/dL; IL-10, in mg/dL
BW | twelve weeks
  body weight, in kg;
BMI | twelve weeks
  body mass index (BMI), in kg/m2, calculated according to weight (kg)/height*height (m)
WC | twelve weeks
  waist circumference, in cm
NC | twelve weeks
  neck circumference, in cm
LAP index | twelve weeks
  Lipid Accumulation Product Index (in cm.mmol.l), calculated for men: men (waist circumference [WC] - 65) x triglycerides (TG), and women (WC - 58) x TG
DAAT index | twelve weeks
  Deep-Abdominal-Adipose-Tissue Index (in cm2), calculated for men (- 382.9 + [1.09 x weight] + [6.04 x waist circumference (WC)] + [- 2.29 x body mass index (BMI)]) and women (- 278 + [- 0.86 x weight] + [5.19 x WC])
VAI index | twelve weeks
  Visceral Adiposity Index (log), calculated for men (waist circumference (WC)/[39 + (1.88 x body mass index (BMI)) x (triglycerides (TG)/1.03) x (1.31/HDL)]) and women (WC/[36.58 + (1.89 x BMI) x (TG/0.81) x (1.53/HDL)])
PFA | twelve weeks
  plasma fatty acids, in percentage
Mon | twelve weeks
  plasma monocytes, in percentage
rs1761667 G>A | baseline
  Polymorphism rs1761667 G>A in the CD36 gene
rs8069645 A>G | baseline
  Polymorphism rs8069645 A>G in the STAT3 gene
Interaction diet * genotype | twelve weeks
  Interaction between dietary intervention, rs1761667 and rs8069645

CONTACTS AND LOCATIONS:
Overall Officials: Aline Marcadenti, PhD, Principal Investigator — Instituto de Cardiologia/Fundação Universitária de Cardiologia (IC/FUC); Vera L Portal, PhD, Study Director — Instituto de Cardiologia/Fundação Universitária de Cardiologia (IC/FUC); Melissa M Markoski, PhD, Study Director — Instituto de Cardiologia/Fundação Universitária de Cardiologia; Alexandre S Quadros, PhD, Study Director — Instituto de Cardiologia/Fundação Universitária de Cardiologia
Locations (1):
- Instituto de Cardiologia/Fundação Universitária de Cardiologia (IC/FUC), Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Dos Santos JL, Portal VL, Markoski MM, de Quadros AS, Bersch-Ferreira A, Marcadenti A. Effect of pecan nuts and extra-virgin olive oil on glycemic profile and nontraditional anthropometric indexes in patients with coronary artery disease: a randomized clinical trial. Eur J Clin Nutr. 2022 Jun;76(6):827-834. doi: 10.1038/s41430-021-01045-7. Epub 2021 Nov 22. PMID 34811509
- [Derived] Campos VP, Portal VL, Markoski MM, Quadros AS, Bersch-Ferreira AC, Garavaglia J, Marcadenti A. Effects of a healthy diet enriched or not with pecan nuts or extra-virgin olive oil on the lipid profile of patients with stable coronary artery disease: a randomised clinical trial. J Hum Nutr Diet. 2020 Jun;33(3):439-450. doi: 10.1111/jhn.12727. Epub 2019 Dec 19. PMID 31856379
- [Derived] Portal VL, Markoski MM, Quadros AS, Garofallo S, Santos JL, Oliveira A, Wechenfelder C, Campos VP, Souza PA, Machado L, Marcadenti A. Effect of polymorphisms in the CD36 and STAT3 genes on different dietary interventions among patients with coronary artery disease: study protocol for a randomized controlled trial. Trials. 2016 Sep 5;17(1):437. doi: 10.1186/s13063-016-1564-1. PMID 27596284